CLINICAL TRIAL: NCT04437511
Title: Assessment of Safety, Tolerability, and Efficacy of Donanemab in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of Donanemab (LY3002813) in Participants With Early Alzheimer's Disease (TRAILBLAZER-ALZ 2)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17737; I5T-MC-AACI (Other: Eli Lilly and Company); 2020-000077-25 (EudraCT Number)
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's; Dementia; Cognitive Impairment; Amyloid Plaque
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Plaque, Amyloid | interventions — donanemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donanemab (Experimental): Participants received 700 milligram (mg) Donanemab every 4 weeks (Q4W) x 3 doses, then 1400 mg Q4W given intravenously (IV) for up to 72 weeks
  Interventions: Drug: Donanemab
- Placebo (Placebo Comparator): Participants received placebo given IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donanemab — Given IV
  Other Names: LY3002813
  Arms: Donanemab
Drug: Placebo — Given IV
  Arms: Placebo

SUMMARY:
The reason for this study is to see how safe and effective the study drug donanemab is in participants with early Alzheimer's disease.

Additional participants will be enrolled to an addendum safety cohort. The participants will be administered open-label donanemab.

Trial participants who were dosed with donanemab in the main study will be enrolled to a 3-year follow up addendum. No study drug will be administered during this follow up.

DETAILED DESCRIPTION:
TRAILBLAZER-ALZ 2 is a Phase 3, double-blind, placebo-controlled study to evaluate the safety and efficacy of N3pG antibody (donanemab) in participants with early symptomatic AD (prodromal AD and mild dementia due to AD) with the presence of brain amyloid and tau pathology.

Following the double-blind 76-week main study period, a double-blind 78-week long-term extension period is added to further evaluate donanemab efficacy and safety over time. Participants from the addendum safety cohort are not eligible for the extension period.

Participants previously dosed with donanemab in the main study will be monitored to track re-accumulation of amyloid plaque for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in memory function reported by participants or informants for ≥ 6 months
* MMSE score of 20 to 28 (inclusive) at baseline
* Meet 18F flortaucipir PET scan (central read) criteria - does not apply to safety cohort
* Meet 18F florbetapir PET scan (central read) criteria
* Have a study partner who will provide written informed consent to participate

Exclusion Criteria:

* Contraindication to MRI or PET scans
* Current treatment with immunoglobulin G (IgG) therapy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1736 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2028-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (274):
- United States (185):
  - Gilbert Neurology, Gilbert, Arizona
  - Xenoscience, Phoenix, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Banner Alzheimer's Institute Tucson, Tucson, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Health Initiatives Research, Fayetteville, Arkansas
  - North County Neurology Associates, Carlsbad, California
  - Wr- Pri, Llc, Encino, California
  - Neuro-Pain Medical Center, Fresno, California
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Clinical Research, Irvine, California
  - Kaizen Brain Center, La Jolla, California
  - Senior Clinical Trials, Inc., Laguna Hills, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - USC Keck School of Medicine, Los Angeles, California
  - Clinical Research Institute, Los Angeles, California
  - Neurovations, Napa, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - SC3 Research - Pasadena, Pasadena, California
  - PCND Neurology, Poway, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Pacific Research Network, San Diego, California
  - Sharp Neurocognitive Research Center, San Diego, California
  - UCSF Memory and Aging Center, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Tilda Research, Tustin, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Colorado Neurological Research Center, PC, Denver, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University, Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Research Center for Clinical Studies, Norwalk, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Neurology Offices of South Florida, Boca Raton, Florida
  - SFM Clinical Research, Boca Raton, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Cohen Medical Associates, Delray Beach, Florida
  - Integrity Clinical Research, Doral, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - MD Clinical, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Encore Research Group- Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Accel Research Sites - Lakeland Clinical Research Unit, Lakeland, Florida
  - ClinCloud - Maitland, Maitland, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - Homestead Associates in Research, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Optimus U Corporation, Miami, Florida
  - Miami Jewish health, Miami, Florida
  - Future Care Solution, Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - The Neurology Research Group, Miami, Florida
  - VIN-Victor Faradji, Miami, Florida
  - Mount Sinai Cancer Center, Miami Beach, Florida
  - Goji Group - Research Trials Group, Miami Lakes, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Synexus Clinical Research US, Inc., Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Emerald Coast Neurology - Airport Boulevard, Pensacola, Florida
  - Quantum Laboratories Clinical Research, Pompano Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Roskamp Institute Clinical Trials Division, Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Brain Matters Research, Stuart, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research - Winter Park, Winter Park, Florida
  - Gwinnett Research Institute, Buford, Georgia
  - Columbus Memory Center, LLC, Columbus, Georgia
  - NeuroStudies, Decatur, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - AMITA Health - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Advocate Medical Group, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - The University of Kansas - Clinical Research Center, Fairway, Kansas
  - College Park Family Care Center/Multi Specialty Clinical Res, Overland Park, Kansas
  - Cotton O'Neil Clinical Research Center - Central Office, Topeka, Kansas
  - Ascension Via Christi Research, Wichita, Kansas
  - Maine Medical Center-Maine Medical Partners Neurology, Scarborough, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - BTC Network, New Bedford, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Donald S. Marks M.D., P.C., Plymouth, Massachusetts
  - Alzheimers Disease Center, Quincy, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Citizens Memorial Hospital District, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Sharlin Health and Neurology, Ozark, Missouri
  - Arch Clinical Trials, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Neurological Associates Albany, Albany, New York
  - Dent Neurologic Institute, Amherst, New York
  - University at Buffalo - UBMD Neurology, Buffalo, New York
  - Clarity Clinical Research, East Syracuse, New York
  - NYU Langone Health, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - CHS-Behavioral Health Research, Charlotte, North Carolina
  - Guilford Neurologic Associates, Inc, Greensboro, North Carolina
  - AMC Research, Matthews, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Cincinnati Physicians Company, LLC, Dayton, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Central States Research, Tulsa, Oklahoma
  - Summit Headlands, Portland, Oregon
  - Center for Cognitive Health, Portland, Oregon
  - Abington Neurological Associates, Ltd., Abington, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Prism Health Richland Department of Neurology Research, Columbia, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Glenn Biggs Institute for Alzheimers & Neurodegenerative Diseases, San Antonio, Texas
  - The Memory Clinic, Bennington, Vermont
  - Integrated Neurology Services - Falls Church, Arlington, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - University of Washington - Harborview Medical Center, Seattle, Washington
  - Kingfisher Cooperative, Spokane, Washington
  - Universal Research Group, Tacoma, Washington
- Australia (9):
  - Central Coast Neurosciences Research, Erina, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - HammondCare Greenwich Hospital, Sydney, New South Wales
  - KARA Institute for Neurological Diseases, Sydney, New South Wales
  - NeuroCentrix, Carlton, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - HammondCare, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Canada (17):
  - OCT Research ULC, Kelowna, British Columbia
  - True North Clinical Research, Halifax, Nova Scotia
  - True North Clinical Research, New Minas, Nova Scotia
  - SKDS Research Inc., Newmarket, Ontario
  - Ottawa Memory Clinic, Ottawa, Ontario
  - Bruyère Research Institute, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Clinique de la Mémoire de l'Outaouais, Gatineau, Quebec
  - MoCA Research and Innovation Inc., Greenfield Park, Quebec
  - Q&T Research Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
- Czechia (6):
  - Clinline Services, Hostivice, Central Bohemia
  - Brain-Soul Therapy, Kladno, Central Bohemia
  - A-Shine, Pilsen, Plzeň-město
  - Clintrial s.r.o., Prague, Praha 10
  - Neurologická Ambulance - Forbeli, Prague, Praha 6
  - Neuropsychiatrie, Prague, Praha 6
- Japan (31):
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - Inage Neurology and Memory Clinic, Inage, Chiba
  - Matsui e-clinic, Akashi, Hyōgo
  - Himeji Central Hospital Affiliated Clinic, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kakigi Dementia Happiness Clinic, Kobe, Hyōgo
  - Tokyo Medical University Ibaraki Medical Center, Inashiki, Ibaraki
  - Memory Clinic Toride, Toride, Ibaraki
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Oita University Hospital, Yufu, Oita Prefecture
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Honmachi Clinic, Ikeda, Osaka
  - Takatsuki General Hospital, Takatsuki, Osaka
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Moriyama Neuro Center Hospital, Edogawa-ku, Tokyo
  - P-One Clinic, Hachiōji, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Tokyo Metro Bokutoh Hospital, Sumida-ku, Tokyo
  - Hiroshima Neurology Clinic, Hiroshima
  - Koseikai Takeda Hospital, Kyoto
  - Ishikawa Clinic, Kyoto
  - National hospital Organization Utano National Hospital, Kyoto
  - Oita Prefectural Hospital, Ōita
  - Itsuki Hospital, Tokushima
  - Tokyo Asbo Clinic, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Makita General Hospital, Tokyo
- Netherlands (4):
  - Brain Research Center Den Bosch B.V., 's-Hertogenbosch, North Brabant
  - Brain Research Center, Amsterdam, North Holland
  - Brain Research Center Zwolle, Zwolle, Overijssel
  - QPS Netherlands B.V, Leeuwarden, Provincie Friesland
- Poland (14):
  - Nzoz Neuro-Kard Ilkowski i Partnerzy SPL, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne NEUROMED, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Ośrodek Badawczo Naukowo Dydaktyczny Chorób Otępiennych Im Księdza Henryka Kardynała Gulbinowicza Uniwersy -T, Ścinawa, Lower Silesian Voivodeship
  - Wroclawskie Centrum Alzheimerowskie, Wroclaw, Lower Silesian Voivodeship
  - Private Practice - Dr. Urszula Chyrchel- Paszkiewicz, Lublin, Lublin Voivodeship
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - Centrum Medyczne NeuroProtect, Warsawawa, Masovian Voivodeship
  - KLIMED Marek Klimkiewicz, Bialystok, Podlaskie Voivodeship
  - Podlaskie Centrum Psychogeriatrii, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne SENIOR, Sopot, Pomeranian Voivodeship
  - Klinika Neuro-Care, Katowice, Silesian Voivodeship
  - Centrum Medyczne Euromedis, Szczecin, West Pomeranian Voivodeship
- Puerto Rico (4):
  - SCB Research Center, Bayamón
  - INSPIRA Clinical Research, San Juan
  - Instituto De Neurologia Dra. Ivonne Fraga, San Juan
  - Barbara Diaz-Hernandez MD Research, Inc., San Juan
- United Kingdom (4):
  - Glasgow Memory Clinic, Motherwell, Great Britain
  - Re:Cognition Health - London, London, London, City of
  - Re:Cognition Health Guildford, Guildford, Surrey
  - Re:Cognition Health - Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Zimmer JA, Sims JR, Evans CD, Nery ESM, Wang H, Wessels AM, Tronchin G, Sato S, Raket LL, Andersen SW, Sapin C, Paget MA, Gueorguieva I, Ardayfio P, Khanna R, Brooks DA, Matthews BR, Mintun MA; Alzheimer's Disease Neuroimaging Initiative. Donanemab in early symptomatic Alzheimer's disease: results from the TRAILBLAZER-ALZ 2 long-term extension. J Prev Alzheimers Dis. 2026 Feb;13(2):100446. doi: 10.1016/j.tjpad.2025.100446. Epub 2025 Dec 1. PMID 41330788
- [Derived] Lu M, Kim MJ, Collins EC, Shcherbinin S, Ellinwood AK, Yokoi Y, Brooks DA, Hansson O, Knopman DS, Sims JR, Mintun MA. Posttreatment Amyloid Levels and Clinical Outcomes Following Donanemab for Early Symptomatic Alzheimer Disease: A Secondary Analysis of the TRAILBLAZER-ALZ 2 Randomized Clinical Trial. JAMA Neurol. 2025 Dec 1;82(12):1251-1256. doi: 10.1001/jamaneurol.2025.3869. PMID 41082199
- [Derived] Chandler JM, Lansdall CJ, Ye W, McDougall F, Belger M, Toth B, Mi X, Sink KM, Atkins AS. The Alzheimer's Disease Cooperative Study - Activities of Daily Living dependence score: revision and validation of an algorithm evaluating patient dependence across the spectrum of AD severity. J Prev Alzheimers Dis. 2025 Sep;12(8):100261. doi: 10.1016/j.tjpad.2025.100261. Epub 2025 Jul 1. PMID 40603145
- [Derived] Zimmer JA, Ardayfio P, Wang H, Khanna R, Evans CD, Lu M, Sparks J, Andersen S, Lauzon S, Nery ESM, Battioui C, Engle SE, Biffi A, Svaldi D, Salloway S, Greenberg SM, Sperling RA, Mintun M, Brooks DA, Sims JR. Amyloid-Related Imaging Abnormalities With Donanemab in Early Symptomatic Alzheimer Disease: Secondary Analysis of the TRAILBLAZER-ALZ and ALZ 2 Randomized Clinical Trials. JAMA Neurol. 2025 May 1;82(5):461-469. doi: 10.1001/jamaneurol.2025.0065. PMID 40063015
- [Derived] Boustani M, Doty EG, Garrison LP Jr, Smolen LJ, Klein TM, Murphy DR, Spargo AW, Belger M, Johnston JA. Estimating the Economically Justifiable Price of Limited-Duration Treatment with Donanemab for Early Symptomatic Alzheimer's Disease in the United States. Neurol Ther. 2024 Dec;13(6):1641-1659. doi: 10.1007/s40120-024-00649-y. Epub 2024 Sep 18. PMID 39292433
- [Derived] Sato S, Hatakeyama N, Fujikoshi S, Katayama S, Katagiri H, Sims JR. Donanemab in Japanese Patients with Early Alzheimer's Disease: Subpopulation Analysis of the TRAILBLAZER-ALZ 2 Randomized Trial. Neurol Ther. 2024 Jun;13(3):677-695. doi: 10.1007/s40120-024-00604-x. Epub 2024 Apr 6. PMID 38581616
- [Derived] Klein EG, Schroeder K, Wessels AM, Phipps A, Japha M, Schilling T, Zimmer JA. How donanemab data address the coverage with evidence development questions. Alzheimers Dement. 2024 Apr;20(4):3127-3140. doi: 10.1002/alz.13700. Epub 2024 Feb 7. PMID 38323738
- [Derived] Sims JR, Zimmer JA, Evans CD, Lu M, Ardayfio P, Sparks J, Wessels AM, Shcherbinin S, Wang H, Monkul Nery ES, Collins EC, Solomon P, Salloway S, Apostolova LG, Hansson O, Ritchie C, Brooks DA, Mintun M, Skovronsky DM; TRAILBLAZER-ALZ 2 Investigators. Donanemab in Early Symptomatic Alzheimer Disease: The TRAILBLAZER-ALZ 2 Randomized Clinical Trial. JAMA. 2023 Aug 8;330(6):512-527. doi: 10.1001/jama.2023.13239. PMID 37459141
- [Derived] Brodtmann A, Darby D, Oboudiyat C, Mahoney CJ, Le Heron C, Panegyres PK, Brew B. Assessing preparedness for Alzheimer disease-modifying therapies in Australasian health care systems. Med J Aust. 2023 Apr 3;218(6):247-249. doi: 10.5694/mja2.51880. Epub 2023 Mar 19. No abstract available. PMID 36934371
- See also: A Study of Donanemab (LY3002813) in Participants with Early Alzheimer's Disease (TRAILBLAZER-ALZ 2) — https://trials.lillytrialguide.com/en-US/trial/4QTyHfYZUZhwbceOEbEqOl

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donanemab | Placebo
Started | 860 | 876
Received at Least One Dose of Drug (Safety Population) | 853 | 874
Completed | 622 | 698
Not Completed | 238 | 178
Not completed — Adverse Event | 50 | 21
Not completed — Death | 15 | 10
Not completed — Lost to Follow-up | 11 | 11
Not completed — Physician Decision | 19 | 10
Not completed — Progressive Disease | 4 | 7
Not completed — Withdrawal by Subject | 111 | 94
Not completed — Withdrawal due to Caregiver Circumstances | 21 | 20
Not completed — Continuing Study | 7 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Donanemab: Participants received 700 mg Donanemab Q4W x 3 doses, then 1400 mg Q4W given IV for up to 72 weeks.
- Total: Total of all reporting groups
Arm/Group | Donanemab | Placebo | Total
Number analyzed (Participants) | 860 | 876 | 1736
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.98 (6.16) | 73.04 (6.20) | 73.01 (6.18)
Sex/Gender, Customized [Number; unit: participants] — Population: Safety Population: All randomized participants who received at least one dose of study drug.
  participants
    Female: number analyzed (Participants) | 853 | 874 | 1727
    Female | 488 | 501 | 989
    Male: number analyzed (Participants) | 853 | 874 | 1727
    Male | 365 | 373 | 738
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 493 | 503 | 996
  Male | 367 | 373 | 740
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 36 | 71
  Not Hispanic or Latino | 583 | 594 | 1177
  Unknown or Not Reported | 242 | 246 | 488
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 57 | 47 | 104
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 21 | 40
  White | 781 | 807 | 1588
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 13 | 4 | 17
  Canada | 64 | 73 | 137
  Czechia | 12 | 10 | 22
  Japan | 45 | 43 | 88
  Netherlands | 13 | 9 | 22
  Poland | 77 | 82 | 159
  United Kingdom | 16 | 23 | 39
  United States | 620 | 632 | 1252
Integrated Alzheimer's Disease Rating Scale (iADRS) [Mean (Standard Deviation); unit: Score on a scale] — Integrated Alzheimer's Disease Rating Scale is used to assess whether donanemab slows down the clinical decline associated with Alzheimer's disease (AD) compared with placebo. iADRS is an integrated assessment of cognition and daily function comprised of items from the Alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance.
  Score on a scale | 104.10 (14.30) | 103.56 (14.02) | 103.83 (14.16)
Screening Tau Category [Count of Participants; unit: Participants] — Population: All randomized participants (pts) who have only evaluable Screening Tau category data.Intermediate tau (Low-medium):All pts with baseline composite tau PET standardized uptake value ratio (SUVr) <= 1.46 and a topographic deposition pattern consistent with advanced AD (AD++) or 1.10 <= SUVr <= 1.46 and a topographic deposition pattern consistent with moderate AD (AD+).High tau:All pts with SUVr >1.46 and topographic deposition pattern consistent with either moderate (AD+) or advanced AD (AD++).
  Participants
    Intermediate (Low-medium): number analyzed (Participants) | 859 | 875 | 1734
    Intermediate (Low-medium) | 588 | 594 | 1182
    High: number analyzed (Participants) | 859 | 875 | 1734
    High | 271 | 281 | 552

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) (Overall Population)
Description: Integrated Alzheimer's Disease Rating Scale is used to assess whether donanemab slows down the clinical decline associated with AD compared with placebo. iADRS is an integrated assessment of cognition and daily function comprised of items from the ADAS-Cog13 and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance. Least Squares (LS) Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, baseline tau level, and baseline acetylcholinesterase inhibitor (AchI)/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline iADRS data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 775 | 824
score on a scale | -10.19 (0.53) | -13.11 (0.50)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = 2.92, 95% CI 2-sided [1.508 to 4.331], Standard Error of Mean 0.72

2. Primary Outcome: Change From Baseline on the Integrated Alzheimer's Disease Rating Scale (iADRS) (Intermediate (Low-medium) Tau Population)
Description: Integrated Alzheimer's Disease Rating Scale is used to assess whether donanemab slows down the clinical decline associated with AD compared with placebo. iADRS is an integrated assessment of cognition and daily function comprised of items from the Alzheimer's disease assessment scale-cognitive subscale (ADAS-Cog13) and the Alzheimer's disease cooperative study-instrumental activities of daily living scale (ADCS-iADL). The scale ranges from 0 to 144, where lower scores indicate worse performance and higher score indicates better performance. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline iADRS data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 533 | 560
score on a scale | -6.02 (0.50) | -9.27 (0.49)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = 3.25, 95% CI 2-sided [1.883 to 4.618], Standard Error of Mean 0.70

3. Secondary Outcome: Change From Baseline on the Mini Mental State Examination (MMSE) Score (Overall Population)
Description: MMSE is an instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, baseline tau level, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline MMSE data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 796 | 841
score on a scale | -2.47 (0.14) | -2.94 (0.13)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p = 0.012, Mixed Models Analysis; LS Mean change difference (Final Values) = 0.47, 95% CI 2-sided [0.104 to 0.841], Standard Error of Mean 0.19

4. Secondary Outcome: Change From Baseline on the Mini Mental State Examination (MMSE) Score (Intermediate (Low-medium) Tau Population)
Description: MMSE is an instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30; lower score indicates greater disease severity. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline MMSE data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 549 | 573
score on a scale | -1.61 (0.14) | -2.09 (0.14)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p = 0.016, Mixed Models Analysis; LS Mean change difference (Final Values) = 0.48, 95% CI 2-sided [0.089 to 0.868], Standard Error of Mean 0.20

5. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) (Overall Population)
Description: The ADAS-Cog13 is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS-Cog13 consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, baseline tau level, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline ADAS-Cog13 data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 797 | 841
score on a scale | 5.46 (0.28) | 6.79 (0.27)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p = 0.0006, Mixed Models Analysis; LS Mean change difference (Final Values) = -1.33, 95% CI 2-sided [-2.086 to -0.565], Standard Error of Mean 0.39

6. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog13) (Intermediate (Low-medium) Tau Population)
Description: The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS-cog consists of 13 items assessing areas of cognitive function most typically impaired in AD: orientation, verbal memory, language, praxis, delayed free recall, digit cancellation. The ADAS-Cog13 scale ranges from 0 to 85. Higher scores indicate greater disease severity. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline ADAS-Cog13 data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 550 | 570
score on a scale | 3.17 (0.27) | 4.69 (0.26)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = -1.52, 95% CI 2-sided [-2.250 to -0.794], Standard Error of Mean 0.37

7. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) (Overall Population)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean value was adjusted for treatment, visit, treatment-by-visit interaction, and covariates for baseline score, baseline score-by-visit interaction, age at baseline, baseline tau category, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline CDR-SB data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 794 | 838
score on a scale | 1.72 (0.096) | 2.42 (0.092)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = -0.70, 95% CI 2-sided [-0.95 to -0.45], Standard Error of Mean 0.127

8. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) (Intermediate (Low-medium) Tau Population)
Description: CDR-SB is a semi-structured interview of participants and their caregivers. Participant's cognitive status is rated across 6 domains of functioning, including memory, orientation, judgment/problem solving, community affairs, home/hobbies, and personal care. Severity score assigned for each of 6 domains; Total score (SB) ranges from 0 to 18. Higher scores indicate greater disease severity. LS Mean value was adjusted for treatment, visit, treatment-by-visit interaction, and covariates for baseline score, baseline score-by-visit interaction, age at baseline, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with baseline Intermediate Tau level and with baseline and at least one postbaseline CDR-SB data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 546 | 569
score on a scale | 1.20 (0.105) | 1.88 (0.102)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = -0.67, 95% CI 2-sided [-0.95 to -0.40], Standard Error of Mean 0.141

9. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study - Instrumental Activities of Daily Living (ADCS-iADL) Score (Overall Population)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities (instrumental activity items 6a, 7-23) of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, baseline tau level, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline ADCS-iADL data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 780 | 826
score on a scale | -4.42 (0.32) | -6.13 (0.30)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p = 0.0001, Mixed Models Analysis; LS Mean change difference (Final Values) = 1.70, 95% CI 2-sided [0.840 to 2.566], Standard Error of Mean 0.44

10. Secondary Outcome: Change From Baseline on the Alzheimer's Disease Cooperative Study - Instrumental Activities of Daily Living (ADCS-iADL) Score (Intermediate (Low-medium) Tau Population)
Description: The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities (instrumental activity items 6a, 7-23) of daily living by participants. The range for the ADCS-iADL is 0-59 with higher scores reflecting better performance. LS Mean value was adjusted for basis expansion terms (two terms), basis expansion term-by-treatment interaction, and covariates for age at baseline, pooled investigator, and baseline AchI/Memantine use.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline Intermediate Tau level and with baseline and at least one postbaseline ADCS-iADL data point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 535 | 562
score on a scale | -2.76 (0.34) | -4.59 (0.32)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = 1.83, 95% CI 2-sided [0.913 to 2.748], Standard Error of Mean 0.47

11. Secondary Outcome: Change From Baseline in Brain Amyloid Plaque Deposition as Measured by Amyloid Positron Emission Tomography (PET) Scan
Description: Amyloid PET scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in amyloid plaques. Quantitative amyloid burden was first formalized as the average Standardized Uptake Value Ratio (SUVR) in six predetermined cortical brain regions relative to the cerebellum as a reference region. Larger SUVR reflects the larger cortical amyloid burden relative to cerebellum. SUVR values were further calibrated to a centiloid (CL) scale. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. LS Mean value was adjusted for treatment, visit, treatment-by-visit interaction, and covariates for baseline score, baseline score-by-visit interaction, baseline tau category, and age at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline amyloid PET scan data point.
Measure: Least Squares Mean (Standard Error); unit: centiloids
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 765 | 812
centiloids | -87.03 (0.950) | -0.67 (0.909)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean change difference (Final Values) = -86.37, 95% CI 2-sided [-88.87 to -83.87], Standard Error of Mean 1.275

12. Secondary Outcome: Change From Baseline in Brain Tau Deposition as Measured by Flortaucipir F18 PET Scan
Description: Flortaucipir PET imaging was used as a quantitative tau biomarker. Tau PET scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in aggregated tau neurofibrillary tangles (NFTs). Quantitative tau burden was formalized using Standardized Uptake Value Ratio (SUVR) in frontal lobe relative to the cerebellum gray as a reference region. Larger SUVR reflects larger tau burden in the frontal lobe relative to cerebellum gray. LS Mean value was adjusted for baseline score, screening tau category, age and treatment (Type III sum of squares).
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and post-baseline tau PET scan.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVR)
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 578 | 654
standardized uptake value ratio (SUVR) | 0.0401 (0.00398) | 0.0442 (0.00374)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Test type: Superiority; p = 0.4522, ANCOVA; LS Mean change difference (Final Values) = -0.0041, 95% CI 2-sided [-0.0148 to 0.0066]

13. Secondary Outcome: Change From Baseline in Brain Volume as Measured by Volumetric Magnetic Resonance Imaging (vMRI)
Description: MRI scans at baseline and at 76 weeks after the first treatment were used to quantitatively estimate change in brain volume. Volumetric MRI parameters were measured in bilateral hippocampus, bilateral whole brain, and bilateral ventricles. LS Mean value was adjusted for treatment, visit, treatment-by-visit interaction, and covariates for baseline score, baseline tau category, and age at baseline.
Time Frame: Baseline, Week 76
Population: All randomized participants with a baseline and at least one postbaseline vMRI data point.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 786 | 831
cubic centimeter (cm^3)
  Bilateral Hippocampus | -0.20 (0.005) | -0.22 (0.005)
  Bilateral Whole Brain | -27.46 (0.409) | -20.79 (0.392)
  Bilateral Ventricles | 10.07 (0.185) | 7.05 (0.178)
Statistical Analysis 1: Comparison: Donanemab vs Placebo; Bilateral Hippocampus; Test type: Superiority; p = 0.002, Mixed Models Analysis; LS Mean change difference (Final Values) = 0.02, 95% CI 2-sided [0.01 to 0.04], Standard Error of Mean 0.007
Statistical Analysis 2: Comparison: Donanemab vs Placebo; Bilateral Whole Brain; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = -6.66, 95% CI 2-sided [-7.76 to -5.56], Standard Error of Mean 0.561
Statistical Analysis 3: Comparison: Donanemab vs Placebo; Bilateral Ventricles; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean change difference (Final Values) = 3.02, 95% CI 2-sided [2.52 to 3.52], Standard Error of Mean 0.256

14. Secondary Outcome: Pharmacokinetics (PK): Average Serum Concentration at Steady State of Donanemab
Description: The average serum concentration at steady state, calculated as Cav = AUCtau/tau, where tau is the dosing interval (4 weeks). AUCtau/tau was assessed at week 12, 16, 24, 36, 52, 64 and Cav for the dosing interval from week 16 to week 20 is reported.
Time Frame: Week 16 to week 20
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Donanemab
Number analyzed (Participants) | 853
micrograms per milliliter (μg/mL) | 63 (32)

15. Secondary Outcome: Number or Participants With Anti-Donanemab Antibodies
Description: Number of participants with treatment-emergent positive Anti-Donanemab antibodies was summarized by treatment group.
Time Frame: Baseline through Week 76
Population: All randomized participants who received at least one dose of study drug and had evaluable anti-drug antibody measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Donanemab | Placebo
Number analyzed (Participants) | 793 | 821
Participants | 693 | 48

ADVERSE EVENTS:
Time Frame: Baseline Up To 76 Weeks plus 57 Days (Follow-up period)
Description: Safety Population: All randomized participants who received at least one dose of study drug. There were 25 deaths reported in subject disposition and 26 deaths in All-cause mortality, because 1 participant death occurred in the plus 57-day follow-up period was considered as completer in the study disposition period. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Donanemab | Placebo
All-Cause Mortality (participants affected / at risk) | 16/853 | 10/874
Serious Adverse Events (participants affected / at risk) | 148/853 | 138/874
Other Adverse Events (participants affected / at risk) | 567/853 | 425/874
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Donanemab (N=853) | Placebo (N=874)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 3 (3) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 9 (9) | 4 (4)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (6) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (2)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (5)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/488 (0) | 1/501 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/488 (1) | 0/501 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metaplastic breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/488 (0) | 1/501 (1)
Mucinous breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/365 (2) | 1/373 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 4 (4) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 13 (13) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (3) | 1 (1)
Syncope (Nervous system disorders) | 9 (9) | 13 (13)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 4 (4) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 3 (3) | 3 (3)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 3 (3)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2/365 (2) | 0/373 (0)
Priapism (Reproductive system and breast disorders) | 1/365 (1) | 0/373 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donanemab (N=853) | Placebo (N=874)
Diarrhoea (Gastrointestinal disorders) | 43 (51) | 50 (56)
Fatigue (General disorders) | 42 (43) | 45 (68)
Covid-19 (Infections and infestations) | 130 (135) | 150 (157)
Urinary tract infection (Infections and infestations) | 42 (52) | 56 (65)
Fall (Injury, poisoning and procedural complications) | 111 (149) | 109 (141)
Infusion related reaction (Injury, poisoning and procedural complications) | 73 (166) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (55) | 41 (44)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 166 (225) | 65 (77)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 200 (270) | 17 (17)
Dizziness (Nervous system disorders) | 52 (59) | 48 (60)
Headache (Nervous system disorders) | 119 (188) | 86 (105)
Superficial siderosis of central nervous system (Nervous system disorders) | 58 (84) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT04437511/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04437511/SAP_001.pdf